CLINICAL TRIAL: NCT02844699
Title: A Multicenter Randomized Double-blind Placebo-controlled Pilot Study of Safety, Pharmacodynamics and Efficacy of Different Treatments of Immunotherapeutic Drug Mobilan (M-VM3) in Patients With Diagnosed Prostate Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Panacela Labs LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PNC-M-VM3-02
Record Dates: First submitted 2016-07-14; First posted 2016-07-26 (Estimated); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; adenovirus; TLR5; immunotherapy; Ad5
MeSH Terms: conditions — Prostatic Neoplasms; Adenoviridae Infections; Alzheimer Disease 5

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mobilan (M-VM3) on both Day 1 and on Day 15 (Experimental): Patients with histologically verified non-metastatic prostate cancer (stage 1 or 3) treated with Investigational Drug Product (Mobilan (M-VM3)) administered 2 weeks apart. All subjects will subsequently undergo planned prostatectomy, ideally within 2 weeks following the final study drug injection and will remain under observation thereafter.
  Interventions: Drug: Mobilan (M-VM3)
- Placebo on Day 1 and Mobilan (M-VM3) on Day 15 (Experimental): Patients with histologically verified non-metastatic prostate cancer (stage 1 or 3) treated with Placebo (Glucose 5%) first on Day 1 and Investigational Drug Product (Mobilan (M-VM3)) in two weeks on Day 15. All subjects will subsequently undergo planned prostatectomy, ideally within 2 weeks following the final study drug injection and will remain under observation thereafter.
  Interventions: Drug: Mobilan (M-VM3); Drug: Placebo
- Placebo on both Day 1 and Day 15 (Placebo Comparator): Patients with histologically verified non-metastatic prostate cancer (stage 1 or 3) treated with Placebo (Glucose 5%) administered 2 weeks apart. All subjects will subsequently undergo planned prostatectomy, ideally within 2 weeks following the final study drug injection and will remain under observation thereafter.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mobilan (M-VM3) — Mobilan (M-VM3), innovative experimental drug based on non-replicate adenoviral delivery system consisting genomic vector coding TLR5-receptor and its ligand 502s.
  Arms: Mobilan (M-VM3) on both Day 1 and on Day 15; Placebo on Day 1 and Mobilan (M-VM3) on Day 15
Drug: Placebo — 5% infusion solution of dextrose (glucose)
  Other Names: Dextrose 5%; Glucose 5%
  Arms: Placebo on Day 1 and Mobilan (M-VM3) on Day 15; Placebo on both Day 1 and Day 15

SUMMARY:
A Phase Ib2, multicenter, randomized, double-blind, placebo-controlled safety and efficacy study evaluating different regimens of the immunotherapeutic drug, Mobilan (M-VM3), in patients with prostate cancer.

DETAILED DESCRIPTION:
Mobilan is a nanoparticle-formulated, recombinant non-replicating adenovirus immunotherapeutic drug that directs expression of both toll-like receptor 5 (TLR5) and a specific agonistic ligand, entolimod (which is a recombinant form of the natural TLR5 ligand, flagellin).

The viral construct infects cells expressing the Coxsackie virus and adenovirus receptor (CAR), which has been shown in preclinical studies to be highly expressed in human prostatic tissue, including prostate cancer tissue. Upon infection, co-expression of both receptor and ligand in the same transfected cell triggers persistent autocrine stimulation of the nuclear factor-kappa B (NF-κB) signaling cascade. In a syngeneic mouse prostate cancer model, prostatic injection of Mobilan leads to activation of an innate immune response with infiltration of neutrophils and natural killer cells (NK) cells and induction of an adaptive immune response, comprising cytotoxic (cluster of differentiation [CD]8+) T cells. Necrotic changes in tumor cells were observed in Mobilan-treated animals with concomitant reductions in prostatic volume. Mobilan also show anti-metastatic activity in a surgical adjuvant mouse model of prostate cancer.

This clinical trial is a Phase Ib double-blinded, randomized, placebo-controlled trial evaluating the efficacy, safety, and pharmacology of either 1 or 2 injections of Mobilan or placebo when administered as neoadjuvant therapy directly into the prostates of patients with newly diagnosed prostate cancer.

All study subjects will receive 2 study drug injections administered 2 weeks apart and will be randomly allocated in a 1:1:1 ratio to 1 of the following 3 drug administration schedules:

* Arm A: Mobilan on both Day 1 and on Day 15.
* Arm B: Placebo on Day 1 and Mobilan on Day 15.
* Arm C: Placebo on both Day 1 and Day 15 Subjects will subsequently undergo planned prostatectomy, ideally within 2 weeks following the final study drug injection and will remain under observation thereafter.

ELIGIBILITY:
Inclusion Criteria:

1. Subscribed Informed consent for participation in the trial
2. Men aged 45 to 75 years
3. Patients with histologically verified prostate cancer, stage Т1-Т3, N0, M0
4. Patient's ECOG status 0-2
5. Negative tests for serologic markers of HIV-infection, viral hepatitis В and С, syphilis
6. Patient and his partner should agree to use barrier contraception throughout the study period

Exclusion Criteria:

1. Failure to obtain Informed consent
2. Clinical or radiological signs of metastases
3. Indication to hormone therapy of prostate cancer
4. Clinically significant cardiovascular diseases:

   * Myocardial infarction within 6 months prior the screening
   * Unstable stenocardia within 3 months prior the screening
   * Severe circulation failure (FC III)
   * Clinically significant arrhythmias
   * Hypotension (systolic blood pressure < 86 mm Hg) or bradycardia with HR < 50 beats per min.
   * Uncontrolled arterial hypertension (systolic blood pressure > 170 mm Hg or diastolic blood pressure > 105 mm Hg.)
5. Clinically significant CNS diseases at the screening
6. Current infection or another severe or systemic disease which increases risk of treatment sequel
7. Pituitary gland or adrenal disorders in medical history
8. Other malignant tumors within the last 5 years
9. Other concomitant diseases in medical history which according to Investigator may aggravate during the study, including uncontrolled diabetes mellitus, rectal diseases, rectal fissures, hemorrhoid, rectal polyps, rectostenosis, inflammatory urinary diseases: chronic prostatitis, cystitis, urethral catheter, chronic urine retention.
10. Complicated allergic history, systemic allergic reaction, any dietary allergy, intolerability, limitations or specific diets which according to the Investigator may be a contraindication for subject participation in the present study.
11. Administration of drug products which have a marked effect on immune system within 3 previous months prior the screening, long-term intake of disaggregants (warfarin, low molecular heparin except for ThromboASS).
12. Participation in other clinical studies or administration of investigational drug products within 30 days prior the screening, or persisting adverse reactions of any investigational drug product.
13. Any clinically significant patient's health disorders and/or laboratory abnormalities not enlisted in the Protocol which are identified at the screening, and/or any reason which according to the Investigator may prevent the patient's participation in the study.
14. Drug or alcohol abuse at the screening or in the past which according to the Investigator makes the patient ineligible for participation in the study.
15. Vaccination made 14 days prior the study
16. Unability to understand or follow study instructions
17. Lack of availability during 6 months after administration of the investigational drug product, fails to follow visit schedule

19. Individual intolerability of the investigational drug product components

Study withdrawal criteria:

1. Any patient may refuse from the study participation on his own wish in any moment on any study stage.
2. Principal Investigator may withdraw any patient from the study in the following cases:

   * Investigator makes the decision that a patient should be withdrawn in his own best interests
   * Patient develops any serious adverse reactions/events in the screening period
   * Patient has been enrolled to the study with violations, or does not follow the protocol requirements
   * Patient needs additional treatment in the screening period
3. Sponsor has right to terminate the study in any moment.
4. Regulatory authorities have right to terminate the study in any moment.

Ages: 45 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2016-07; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Frequency and intensity of adverse events (according to CTCAE v 4.03 classification) | Baseline to up to 45 days after the first drug administration
Counting of CD4+ and CD8+ cells in prostate biopsy and surgery samples | Baseline to up to 45 days after the first drug administration
  Using immunological assays

SECONDARY OUTCOMES:
Change in total Prostate-specific antigen (PSA) level | Baseline to up to 45 days after the first drug administration
Value of the Irani score of post-operative prostate tissue (if material is available for analysis) | On Day 30 after the first drug administration
  Irani J (1997) scale include histological assessment of slide mounts obtained after operation as follow:
  Degree of immune cell infiltration:
  0 - No inflammatory cells, 1 - Scattered inflammatory cell infiltrate within the stroma without lymphoid nodules, 2 - Nonconfluent lymphoid nodules, 3 - Large inflammatory areas with confluence of infiltrate
Value of the Gleason score of post-operative prostate tissue (if material is available for analysis) | On Day 30 after the first drug administration
  The Gleason grading system is used to evaluate the stage of prostate cancer using samples from biopsy or post- surgical samples as follow:
  1 - The cancerous prostate closely resembles normal prostate tissue. 2 - The tissue still has well-formed glands, but they are larger and have more tissue between them. 3 - The tissue still has recognizable glands, but the cells are darker. 4 - The tissue has few recognizable glands. 5 - The tissue does not have any or only a few recognizable glands.
Plasma concentration of inflammatory cytokines | Baseline to up to 45 days after the first drug administration
Presence of protein 502s in blood plasma | Baseline to up to 45 days after the first drug administration
  Using ELISA assay
Presence of protein 502s in prostate biopsy and surgery samples | Baseline to up to 45 days after the first drug administration
  Using ELISA assay
Presence of protein TLR5 in prostate biopsy and surgery samples | Baseline to up to 45 days after the first drug administration
  Using ELISA assay

CONTACTS AND LOCATIONS:
Locations (4):
- Russia (4):
  - Moscow State Budgetary Healthcare Institution "City Clinical Hospital № 57" of Moscow Healthcare Department, Moscow
  - Moscow State University of Medicine and Dentistry, Moscow
  - Federal State Budgetary Institution "Saint Petersburg Clinical Scientific and Practical Center for Special types of medical care (Oncological)", Saint Petersburg
  - Federal State Budgetary Institution "Scientific Research Oncology Institute named after N.N. Petrov" of the Ministry of Health of the Russian Federation, Saint Petersburg